CLINICAL TRIAL: NCT02867683
Title: The Effects of Vibrotactile Feedback During Vestibular Rehabilitation
Brief Title: Vibrotactile Feedback During Vestibular Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Michigan (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Susan Whitney, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO13020399; 5R21DC012410 (NIH)
Record Dates: First submitted 2016-08-04; First posted 2016-08-16 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Vestibular Disease
Keywords: vibrotactile feedback; vestibular rehabilitation; balance
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vibrotactile Feedback (Experimental): Balance exercises completed while vibration was applied to the trunk (anterior, posterior, right, and left) if postural sway exceeded a pre-determined threshold during the exercise.
  Interventions: Other: Vibrotactile Feedback
- Without Vibrotactile Feedback (No Intervention): Balance training without feedback

INTERVENTIONS:
Other: Vibrotactile Feedback — Balance training Vibrotactile feedback applied to the trunk
  Arms: Vibrotactile Feedback

SUMMARY:
This study evaluates the use of vibrotactile feedback to traditional vestibular treatment protocols. Half the patients will have vibrotactile feedback added to their treatment protocols while the other half will undergo traditional vestibular treatment without vibrotactile feedback.

DETAILED DESCRIPTION:
Vestibular and balance rehabilitation is an effective way to improve balance for individuals with balance impairments by using the strategies of adaptation, habituation, or substitution. Typical vestibular treatment is usually 3 sessions per week for 6 weeks. For people with uncompensated unilateral vestibular hypofunction or bilateral vestibular loss, recovery/adaptation is often incomplete and chronic balance impairments result.

Vibrotactile feedback (VTF) is a strategy of substitution, or augmentation, to replace disrupted or absent vestibular function. The sensory information replaces disrupted or absent vestibular function to give persons additional signals about their body position in space. Real-time VTF applied to the trunk has been shown to decrease postural sway but the long-term benefits of training with VTF on balance and function have not been examined.

ELIGIBILITY:
Inclusion Criteria:

* unilateral peripheral vestibular hypofunction
* bilateral peripheral vestibular hypofunction

Exclusion Criteria:

* confounding neurologic or neuromuscular disorders
* pregnancy
* inability to stand for 3 minutes
* recent lower extremity fracture/severe sprain within the last 6 months
* previous lower extremity joint replacement
* incapacitating back or lower extremity pain
* body too large for equipment

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-10; Primary Completion 2017-08-01 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Sensory Organization Testing | Baseline, 3 weeks, 6 weeks, 10 weeks, & 30 weeks
  Postural sway data will be collected during Computerized Dynamic Posturography using the NeuroCom Equitest.
Change in 10-meter walk test | Baseline, 3 weeks, 6 weeks, 10 weeks, & 30 weeks
  Participants preferred gait velocity will be assessed while walking in a straight path by timing 10-meter walk.
Change in Dynamic Gait Index and Functional Gait Assessment | Baseline, 3 weeks, 6 weeks, 10 weeks, & 30 weeks
  Measures that assess ability to modify walking in the presence of external demands. Includes tasks such walking with head turns, walking around obstacles, stepping over obstacles, and negotiating stairs. Each task is scored on a 4 point scale (0-3) and a total score is compiled.
Change in Five Times Sit to Stand | Baseline, 3 weeks, 6 weeks, 10 weeks, & 30 weeks
  A stopwatch is used to record the amount of time it takes the participant to move from a seated position to a standing position back to seated without using their hads for a total of 5 repetitions

SECONDARY OUTCOMES:
Change in Activities-specific Balance Confidence Scale | Baseline, 3 weeks, 6 weeks, 10 weeks, & 30 weeks
  A 16-item self-report instrument which the participants completes by scoring their perceived confidence level during activities of daily living.
Change in Dizziness Handicap Inventory | Baseline, 3 weeks, 6 weeks, 10 weeks, & 30 weeks
  A self-report instrument which the participants indicates whether or not the listed 25 activities cause dizziness.
Change in Short Form-12 | Baseline, 3 weeks, 6 weeks, 10 weeks, & 30 weeks
  A 12 question self-report instrument that provide information about mental and physical functioning as well as health-related quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided